CLINICAL TRIAL: NCT07117812
Title: Feasibility and Safety of Laparoscopic Purse-string Suture Clamp and Multi-functional Seal Cap for Totally Laparoscopic Radical Total Gastrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Li Yang, Prof., The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-SR-633
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Gastric Cancer (GC); Gastrectomy; Anastomosis, Roux-en-Y; Laparoscopic
MeSH Terms: conditions — Stomach Neoplasms | interventions — methionine synthase reductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic Roux-en-Y esophagojejunostomy using purse-string forceps and sealing ring (Experimental): Performing totally laparoscopic radical total gastrectomy with R0 resection, completing esophagojejunostomy using purse-string forceps and multifunctional sealing ring.
  Interventions: Procedure: Laparoscopic purse-string forceps and multifunctional sealing ring

INTERVENTIONS:
Procedure: Laparoscopic purse-string forceps and multifunctional sealing ring — Performing totally laparoscopic radical total gastrectomy with R0 resection, completing esophagojejunostomy using purse-string forceps and multifunctional sealing ring.
  Other Names: LPSF and MSR

SUMMARY:
Currently, there are three main methods for endoscopic esophagojejunostomy: circular, linear, and hand-sewn anastomosis, but no universally accepted optimal approach has been established.

Hand-sewn anastomosis relies on advanced endoscopic suturing skills, making it technically demanding and only performed in a limited number of hospitals.

Linear anastomosis is simple to perform and the most widely used in clinical practice. However, it requires resection of a longer segment of the distal esophagus and may struggle to ensure adequate margins for high-positioned tumors or unclear resection boundaries.

Circular anastomosis is a classic method. Its end-to-side approach preserves more esophageal length, making it suitable for high-positioned tumors without the need to close a common opening. Various techniques (e.g., the reverse-puncture method and the Orvil™ transoral anvil technique) have been reported. However, due to challenges such as purse-string suturing, complex anvil placement, and restricted stapler maneuverability, widespread adoption remains difficult.

Prof. Du Jianjun's team innovatively employed endoscopic purse-string forceps and a multifunctional sealing ring to achieve circular anastomosis, demonstrating preliminary technical advantages. This study further explores its feasibility and short-term outcomes in totally endoscopic total gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years, regardless of gender; Histologically confirmed gastric or gastroesophageal junction (GEJ) adenocarcinoma. For GEJ cancer, only Siewert type III and type II (without requiring thoracotomy) are eligible (applicable to multiple primary cancers); Preoperative assessment by a gastrointestinal surgeon and imaging specialist confirming cStage I-III disease with eligibility for curative-intent R0 resection. Patient consents to surgery and is deemed surgically fit by the surgeon; Anticipated R0 resection achievable via total gastrectomy with D1+/D2 lymphadenectomy; Expected survival ≥6 months; ECOG Performance Status (PS) score (see Appendix 2) of 0 or 1; Adequate major organ function; Body weight ≥40 kg or BMI >18.5 and <30 kg/m²; No prior chemotherapy, radiotherapy, targeted therapy, or immunotherapy; Patient has read and fully understood the informed consent form and voluntarily signed it

Exclusion Criteria:

* History of other active malignancies within the past 5 years or concurrent malignancies (except cured localized tumors such as basal cell carcinoma, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate/cervix/breast, Stage I lung/colorectal cancer, etc.).

Previous upper abdominal surgery (excluding laparoscopic cholecystectomy). History of gastrectomy, endoscopic mucosal resection (EMR), or endoscopic submucosal dissection (ESD).

Requirement for concurrent surgery for other diseases. Emergency surgery due to gastric cancer complications (bleeding, obstruction, or perforation).

Planned or prior organ/bone marrow transplantation. Blood transfusion within 2 weeks before surgery, bleeding history, or Grade ≥3 hemorrhage (CTCAE v4.0) within 4 weeks.

Coagulopathy (INR >1.5 without anticoagulants) or use of anticoagulants (warfarin/heparin). Prophylactic low-dose warfarin (≤1 mg/day) or aspirin (≤100 mg/day) is permitted if INR ≤1.5.

Arterial/venous thrombosis within 6 months (e.g., stroke, DVT, pulmonary embolism), excluding catheter-related thrombosis from prior chemotherapy.

Myocardial infarction within 6 months or uncontrolled arrhythmia (QTc ≥450 ms [men]/≥470 ms [women] by Fridericia's formula).

NYHA Class III-IV heart failure or LVEF <50%. Ventilatory dysfunction (FEV1 <50% predicted). Urinary protein ≥++ or 24-hour urine protein >1.0 g. Clinically significant pleural/peritoneal effusion requiring intervention. HIV infection. Active tuberculosis. Non-healing wounds or incomplete fracture healing. Active/suspected autoimmune disease (stable cases without immunosuppressants allowed).

Severe autoimmune diseases (e.g., SLE, IBD), chronic diarrhea disorders, or active HBV/HCV (HBV DNA <500 copies/mL permitted).

Systemic corticosteroids (>10 mg/day prednisone equivalent) within 14 days (topical/inhaled steroids or physiologic replacement doses allowed).

Active infection requiring systemic antibiotics within 14 days (prophylactic antibiotics permitted).

Live vaccines within 28 days (inactivated flu vaccines allowed). Concurrent participation in another surgical trial. Alcohol/drug abuse history (abstinent patients eligible). Non-compliance or incomplete data affecting safety/efficacy assessments. Pregnancy/lactation. Other conditions deemed high-risk by investigators. Investigator-determined ineligibility.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Early postoperative complications | 30 days
  Early postoperative complications were defined as adverse events occurring within 30 days after surgery. All complications were classified according to the Clavien-Dindo grading system and recorded numerically.

SECONDARY OUTCOMES:
Postoperative recovery situation | 30 days
  The time of first getting out of bed after surgery, the time of postoperative ventilation, the time of liquid diet after surgery, the time of soft food after surgery, the length of hospital stay after surgery, and the total amount of abdominal drainage; The changes of albumin, prealbumin, white blood cells, hemoglobin, C-reactive protein, IL-6, etc. in the peripheral blood after surgery.
Late postoperative complications | 2 years
  Events observed from day 31 to month 24 after surgery.

IPD SHARING:
Plan to Share IPD: Undecided